CLINICAL TRIAL: NCT07039383
Title: Kymriah Real-world Effectiveness in ALL (KareALL): a Retrospective Chart Review Study of Tisagenlecleucel-treated ALL Patients
Brief Title: A Real-world Study of the Effectiveness of Tisagenlecleucel in Acute Lymphoblastic Leukemia Patients
Acronym: KareALL
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CCTL019BUS08
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Tisagenlecleucel; Real-world; Chart review
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Tisa-cel Cohort: Patients with R/R B-cell ALL who received tisa-cel infusions between December 2020 and September 2022.

SUMMARY:
This was a retrospective, cross-sectional, center-based chart review study that collected real-world data for relapsed/refractory (R/R) acute lymphoblastic leukemia (ALL) patients receiving tisagenlecleucel (tisa-cel). Five centers in the United States were included for the study.

The date of the initial tisa-cel infusion was defined as the index date. A baseline period from ALL diagnosis to the index date was used to capture patient characteristics including demographics, and disease and treatment history. The study period, defined as the period from tisa-cel infusion to the end of follow-up date, i.e. the last contact date on medical charts or death, whichever was earlier, was used to capture the clinical outcomes of tisa-cel among ALL patients.

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with B-cell ALL.
* Infusion of tisa-cel happened since December 2020 and at least 1 year before the chart abstraction date.

Exclusion criteria: None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Remission Rate | Month 1 and Month 3
  Remission rate was defined as the best overall response as either complete remission (CR) or complete remission with incomplete blood count recovery (CRi) to tisa-cel.
  CR: <5% blasts in bone marrow based on morphologic assessment, no evidence of extramedullary disease, full recovery of peripheral blood counts (platelets > 100x10^9/L, absolute neutrophil > 1.0x10^9/L, and circulating blasts <1%), and blood transfusions independency (i.e., no transfusion or transfusion ≤7 days).
  CRi: <5% blasts in bone marrow, no evidence of extramedullary disease, but without full recovery of peripheral blood counts with or without blood transfusions independency.

SECONDARY OUTCOMES:
Number of Patients per Demographic Category | Baseline
  Demographic categories included:
  * Age group
  * Gender
  * Race
  * Ethnicity
  * Geographical region
  * Distance between residence and referral center (<5, 5-30, 30-60, >60 miles)
  * Type of insurance
Demgraphics: Weight | Baseline
Number of Patients by Disease Characteristics Category | Baseline
  Disease characteristics categories included:
  * Relapse or refractory status before tisa-cel infusion
  * CD19 tumor expression among relapsed patients before tisa-cel infusion
  * Karnofsky or Lansky performance score (PS)
  * Lymphoblast proportion in bone marrow (<5%, >= 5%)
  * Conditions of interest before tisa-cel infusion
  * Patients with relapse before tisa-cel infusion
  * Number and type of relapse before tisa-cel infusion (any bone marrow and/or central nervous system relapse)
  * Cytogenic testing performed at tisa-cel infusion
  * Cytogenic abnormalities at tisa-cel infusion
  * Number of distinct cytogenic abnormalities (1, 2, 3, 4+)
  * Comorbidities at tisa-cel infusion
  * Remission status at time of tisa-cel infusion
  The Karnofsky and Lansky PS are measures of functional impairment. They run from 0 to 100, where 0 is death and 100 is normal health. The Karnofsky scale is for patients aged 16 years or older. The Lansky scale is for patients younger than 16 years old.
Number of Patients by Treatment Characteristics Category | Baseline
  Treatment characteristic categories included:
  * Treatments of interest before tisa-cel infusion
  * Number of prior lines of treatment category (1 to 7)
  * Received prior allogenic stem cell transplant (alloSCT)
  * Number of alloSCT received (0, 1, 2)
  * Year of initial tisa-cel infusion
  * Bridging treatment agent received before tisa-cel infusion
  * Lymphodepleting regimen received before tisa-cel infusion
  * Type of tisa-cel infusion dose received (single, multiple)
  * Weight at tisa-cel infusion (<= 50 kilograms [kg], >50 kg)
Lymphoblast Proportion in Bone Marrow Before Tisa-cel Infusion | Baseline
ALL Disease Duration at Tisa-cel Infusion | Baseline
Time From Initial Diagnosis to First Relapse | From initial diagnosis up to first tisa-cel infusion, approximately 13 years
Number of Patients by Time From Initial Diagnosis to First Relapse | Baseline
  Time intervals: <18 months, 18-36 months, and >36 months.
Time From Most Recent Relapse to Initial Tisa-cel Infusion | From initial diagnosis up to first tisa-cel infusion, approximately 13 years
Number of Lines of Treatment Prior to Tisa-cel Infusion | Baseline
Time From Tisa-cel Infusion to Loss of Follow-up or Death due to Any Cause | Baseline up to approximately 3 years
Time From Leukapheresis to Tisa-cel Infusion | From initial diagnosis up to first tisa-cel infusion, approximately 13 years
Number of Doses for Initial Tisa-cel Infusion | Baseline
  Number of doses for initial infusion was measured among those who received multiple doses.
Weight Adjusted Transduced Cell Dose Infused in Patients Who Weighed 50 kg or Less at Tisa-cel Infusion | Baseline
Total Cell Dose Infused in Patients Who Weighed More Than 50 kg at Tisa-cel Infusion | Baseline
Number of Patients by Conditions Experienced After Tisa-cel Infusion | Baseline up to approximately 3 years
Number of Patients by Bone Marrow Minimal Residual Disease (MRD) Status | Month 1 and Month 3
  Bone marrow MRD is a measure of the number of cancer cells remaining in the body after treatment. The number of patients overall with bone marrow MRD negative and those who achieved CR or CRi response with bone marrow MRD negative after tisa-cel infusion was measured. Bone marrow MRD negative was based on clinical assessment by the investigator.
  CR: <5% blasts in bone marrow based on morphologic assessment, no evidence of extramedullary disease, full recovery of peripheral blood counts (platelets > 100x10^9/L, absolute neutrophil > 1.0x10^9/L, and circulating blasts <1%), and blood transfusions independency (i.e., no transfusion or transfusion ≤7 days).
  CRi: <5% blasts in bone marrow, no evidence of extramedullary disease, but without full recovery of peripheral blood count with or without blood transfusions independency.
Duration of Remission (DOR) | Months 1, 6, 12, 18, 24, and 30
  DOR was defined as the time from onset of remission to relapse or death due to ALL.
  Relapse was defined as:
  * Reappearance of blasts in the blood (≥1%), or
  * Reappearance of blasts in bone marrow (≥5%), or
  * Appearance of any extramedullary disease
Relapse-free Survival (RFS) | Months 1, 6, 12, 18, 24, and 30
  RFS was defined as the time from onset of remission to relapse or death due to any cause.
  Relapse was defined as:
  * Reappearance of blasts in the blood (≥1%), or
  * Reappearance of blasts in bone marrow (≥5%), or
  * Appearance of any extramedullary disease
Event-free Survival (EFS) | Months 1, 6, 12, 18, 24, and 30
  EFS was defined as the time from tisa-cel infusion to the earliest of the following events: death due to any cause, relapse, treatment failure (i.e., no response), or new anticancer therapy for ALL (i.e., treatments other than tisa-cel or SCT).
  Relapse was defined as:
  * Reappearance of blasts in the blood (≥1%), or
  * Reappearance of blasts in bone marrow (≥5%), or
  * Appearance of any extramedullary disease
Overall Survival (OS) | Months 1, 6, 12, 18, 24, and 30
  OS was defined as the time from tisa-cel infusion to the date of death due to any cause.
Number of Patients who had AlloSCT After Tisa-cel Infusion | Up to approximately 3 years
  Patient counts were categorized by:
  * Pre-planned/not pre-planned at time of tisa-cel infusion
  * Achieved/had not achieved B-cell recovery at time of alloSCT
  * Unknown B-cell recovery status
  * Did not have B-cell aplasia
  * alloSCT received within 12 months after tisa-cel infusion
  * Relapse status after tisa-cel infusion before alloSCT
Time From Tisa-cel Infusion to Subsequent AlloSCT | Baseline up to approximately 3 years
Number of Patients by Tisa-cel Reinfusion Received After Initial Infusion | Up to approximately 3 years
  Patient counts were categorized by:
  * Received/did not receive reinfusion
  * Received infusion within 12 months after initial infusion
  * Reason for reinfusion
Time From Initial Tisa-cel Infusion to Tisa-cel Reinfusion | Baseline up to approximately 3 years
Number of Patients by Type of new Anticancer Therapy (Other Than AlloSCT or Reinfusion) Received After Tisa-cel infusion | Up to approximately 3 years
Number of Patients by B-cell Aplasia Status After Tisa-cel Infusion | Up to approximately 3 years
  B-cell aplasia status included:
  * Experienced B-cell aplasia
  * Recovered from B-cell aplasia
Time from Tisa-cel Infusion to B-cell Aplasia | Baseline up to approximately 3 years
Number of Patients by use of Immunoglobulin (Ig) Replacement Therapy Among Those who Experienced B-cell Aplasia | Up to approximately 3 years
  Ig replacement therapy use was categorized as follows:
  * Received Ig replacement therapy
  * Received intravenous immunoglobulin (IVIG) therapy
  * Ongoing IVIG therapy
  * Stopped IVIG therapy
  * Received subcutaneous immunoglobulin (SCIG) therapy
  * Ongoing SCIG therapy
  * B-cell aplasia recovered
Average Dose of Ig Replacement Therapy | Up to approximately 3 years
  Ig replacement therapy included IVIG and SCIG.
Duration of Ig Replacement Therapy | Up to approximately 3 years
  Ig replacement therapy included IVIG and SCIG.
Rate of Maintenance of B-cell Aplasia | Months 1, 2, 3, 6, 9, 12, 18, 24, 30
Number of Patients by Hospitalizations at Initial Tisa-cel Infusion | Baseline
  Hospitalization categories included not hospitalized, hospitalized for Tisa-cel infusion, and subsequently admitted to intensive care unit (ICU).
Length of Stay in Hospital for Initial Tisa-cel Infusion | Up to approximately 3 years
Number of Patients by Hospitalizations After Tisa-cel Infusion | Up to approximately 3 years
  Hospitalization categories included hospitalized, not hospitalized, and first hospitalization.
Number of Hospitalizations After Tisa-cel Infusion | Up to approximately 3 years
Length of Stay in Hospital After Tisa-cel Infusion | Up to approximately 3 years
Time From Initial Tisa-cel Infusion to the First Hospitalization | Baseline up to approximately 3 years
Number of Patients by Primary Reason for the First Hospitalization | Up to approximately 3 years
Number of Patients by ICU Admissions After Tisa-cel Infusion | Up to approximately 3 years
  ICU admission categories included admitted to ICU, not admitted to ICU, and first ICU admission.
Number of ICU Admissions After Tisa-cel Infusion | Up to approximately 3 years
Length of Stay per ICU Admission After Tisa-cel Infusion | Up to approximately 3 years
Number of Patients by Primary Reason for ICU Admission After Tisa-cel Infusion | Up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States